CLINICAL TRIAL: NCT03748628
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]EDP-305 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Absorption, Metabolism and Excretion (AME) Study of [14C]EDP-305 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 305-009
Record Dates: First submitted 2018-10-31; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: AME Study
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — EDP-305

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm EDP-305 (Experimental)
  Interventions: Drug: EDP-305

INTERVENTIONS:
Drug: EDP-305 — [14C]EDP-305

SUMMARY:
A Phase 1, Open-label Study of the absorption, metabolism, and excretion of a single oral dose of [14C]EDP-305 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 18 and 55 years (inclusive) with a body mass index between 18.0 and 32.0 kg/m2 (inclusive)
* able to comprehend and willing to sign an Informed Consent Form
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (including gastrectomy and cholecystectomy; uncomplicated appendectomy and hernia repair will be allowed).
* Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-305 in plasma | Up to 9 days
AUC of EDP-305 in plasma | Up to 9 days
AUC-inf in plasma | Up to 9 days

SECONDARY OUTCOMES:
Amount excreted in urine (Aeu) | Up to 9 days
Amount excreted in feces (Aef) | Up to 9 days
Safety measured by adverse events | Up to 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States